CLINICAL TRIAL: NCT03726203
Title: Benign Gynecologic Laparoscopic Surgery: Comparison of Conventional Trocars to the Teleflex® MiniLap® System in Length of Hospitalization, Pain and Aesthetics, a Randomized Study.
Brief Title: Laparoscopic Surgery: Comparison of Conventional Trocars to the Teleflex® MiniLap® System
Acronym: MiniTroc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Teleflex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017_81; 2018-A01276-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Gynecologic Surgeries
Keywords: Laparoscopy; Trocar; MiniLap; surgery; gynecology; pain, scars; scars
MeSH Terms: conditions — Pain; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trocars of type MiniLap (Experimental): Patients benefiting from the use of trocars of type MiniLap of Teleflex during the realization of their coelioscopy scheduled in ambulatory
  Interventions: Device: laparoscopic gynecologic surgery with the MiniLap System.
- trocars classics (Active Comparator): Patients benefiting from the use of trocats classics during the realization of their coelioscopy scheduled(programmed) in ambulatory.
  Interventions: Device: laparoscopic gynecologic surgery with the conventional single-use trocars.

INTERVENTIONS:
Device: laparoscopic gynecologic surgery with the MiniLap System. — Subjects participating in the study will undergo laparoscopic gynecologic surgery as planned in the routine care, but using the MiniLap System instead of the conventional single-use trocars used usually.
  Arms: trocars of type MiniLap
Device: laparoscopic gynecologic surgery with the conventional single-use trocars. — Subjects participating in the study will undergo laparoscopic gynecologic surgery as planned in the routine care using the conventional single-use trocars used usually.
  Arms: trocars classics

SUMMARY:
During laparoscopy, trocars are essential: they allow the passage of instruments through the wall. In gynecology, with exception, trocars 5mm (used for the passage of endo-scissors and forceps) and 10 to 12mm are used (especially for optics).

Trocars are responsible for complications, such as vascular wounds, digestive wounds, pain, infections or postoperative hernias, or aesthetic sequelae, and should be chosen with caution: most complications of laparoscopy are essentially due to their placement, and the complications at the introduction of the first trocar are the most frequent.

The MiniLap® system developed by Teleflex does not require trocars in the case of a single forceps, or a single 5mm trocar with the necessary forceps change (this is the Percuvance® system). The aim of the latter is to make minimally invasive surgery even less invasive, thanks to a reduction in the number of trocars used (in many cases, elimination of two trocars), smaller incisions (percutaneous use of instruments, with a diameter of 2,4mm) thus reducing the complications

ELIGIBILITY:
Inclusion Criteria:

* BMI <35kg / m2
* No history of multiple abdominopelvic surgery
* Without absolute contraindication to laparoscopy
* In the context of ambulatory surgery
* With precise laparoscopy of indication:

  * Exploratory or diagnostic
  * Exploration of infertility
  * Performing a tubal permeability test
  * Performing a salpingectomy
  * Realization of a tubal sterilization
  * Realization of a tubal plasty
  * Performing an ovariectomy
  * Performing a simple ovarian cystectomy
* Patient have been informed during her preoperative consultation and have signed the consent in a free and informed manner upon admission to hospital

Exclusion Criteria:

* Performing an emergency surgery
* Carcinological surgery
* Performing a benign but complex surgery such as:

  * Hysterectomy
  * Prolapse cure
  * promontofixation
  * Complex surgery of endometriosis
  * Removal of large cyst from the ovary.
* Person unable to receive informed information and / or give consent. Person deprived of liberty.
* Pregnant or nursing woman.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
The time required to validate the Marshall and Chung criteria authorizing outpatient discharge when using the Minilap® system in comparison to the use of conventional trocars. | at the end of surgery, an average 3 hours

SECONDARY OUTCOMES:
Pain using the Visual Analog Scale (VAS) | at immediate postoperative (baseline,1 hour and 3 hours) and postoperative visit (6 weeks ± 1 after surgery).
  subjective evaluation of pain of the patient by 0 to 10 scale
Aesthetic scars using a scale of 0 to 10 | postoperative visit (6 weeks ± 1 after surgery).
  subjective evaluation of the patient and the surgeon by means of a 0 to 10 scale
number of complication per operative | At immediate postoperative (baseline,1 hour and 3 hours)
  collection of the complications per operating by means of a questionnaire to be filled(performed) by the surgeon at the end of intervention
of the intraoperative use of the trocar system using a questionnaire to be completed by the surgeon | At immediate postoperative (baseline,1 hour and 3 hours)
post-operative complications at the level of the trocar apertures using a questionnaire | at immediate postoperative (baseline,1 hour and 3 hours) and postoperative visit (6 weeks ± 1 after surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Chrystelle Rubod, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandres, CHU, Lille, France